CLINICAL TRIAL: NCT04330820
Title: Phase-I/II Trial for Relapsed or Refractory AML Patients Combining Cytarabine and Mitoxantrone With Venetoclax (RELAX)
Brief Title: Trial for Relapsed or Refractory AML Patients Combining Cytarabine and Mitoxantrone With Venetoclax (RELAX)
Acronym: RELAX
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TUD-RELAX1-070
Record Dates: First submitted 2020-03-19; First posted 2020-04-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Relapsed Adult AML; Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: The phase I part will be conducted according to the enhanced algorithms of a 3+3H design (Ji et al. J Clin Oncol 2013).
  The phase II part will be performed as single stage study adopting the A'Hern design (A'Hern Stat Med 2001).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax+Cytarabin+ Mitoxantron (Experimental): The treatment plan combines a fixed dose of venetoclax and mitoxantrone with increasing doses of cytarabine (V-MAC).
  Interventions: Drug: Venetoclax Oral Tablet

INTERVENTIONS:
Drug: Venetoclax Oral Tablet — This study will investigate the combination of a fixed maximum venetoclax dose with increasing cytarabine doses plus mitoxantrone in a fixed dose in phase I. In Phase II cytarabine will be given at MDT or RP2D that assessed in phase I.
  The venetoclax dose of 400 mg will be reached by a ramp up over 3 days. Parallel chemotherapy with cytarabine and mitoxantrone will start on day 3.
  Other Names: Cytarabin

SUMMARY:
This is an open-label Phase I dose-escalation study of oral venetoclax in combination with increasing cytarabine doses plus mitoxantrone to define the safety profile and MTD of cytarabine in subjects with a histologically or cytologically confirmed acute myeloid leukemia who are refractory or suffered a relapse. This study will be conducted at multiple centers in Germany.

DETAILED DESCRIPTION:
* To determine safety, tolerability, maximum tolerated dose, and recommended phase II dose of venetoclax in combination with increasing cytarabine doses plus fixed dose mitoxantrone in subjects with a relapsed or refractory AML considered fit for intensive salvage therapy.
* To assess the preliminary efficacy of venetoclax in combination with increasing cytarabine doses plus fixed dose mitoxantrone in subjects with a relapsed or refractory AML considered fit for intensive salvage therapy.

ELIGIBILITY:
Inclusion criteria for both escalation and expansion phase:

* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained before screening.
* AML according to WHO-2016 criteria, excluding acute promyelocytic leukemia
* Relapsed from first or second CR after 1-2 cycles of standard induction chemotherapy (which must have included cytarabine with an anthracycline or anthracenedione), including relapse after allogeneic stem cell transplantation (dose escalation and expansion part)
* Age 18-75 years
* Fit for intensive chemotherapy, defined by

  * ECOG 0-2, life expectancy > 3months
  * Adequate hepatic function: ALAT/ASAT/Bilirubin ≤2.5 x ULN*

    * unless considered due to leukemic organ involvement Note: Subjects with Gilbert's Syndrome may have a bilirubin > 2.5 × ULN per discussion between the investigator and Coordinating investigator.
  * Adequate renal function assessed by serum creatinine ≤ 1.5x ULN OR creatinine clearance (by Cockcroft Gault formula) ≥ 50 mL/min
* Patient is afebrile and hemodynamically stable for at least 72 hours at the time of study medication initiation.
* Male subjects must agree to refrain from unprotected sex and sperm donation from time point of signing the informed consent until 30 days after the last dose of study drug.
* Women must fulfill at least one of the following criteria in order to be eligible for trial inclusion:

  * Post-menopausal (12 months of natural amenorrhea or 6 months of amenorrhea with Serum FSH > 40 U/ml)
  * Postoperative (i.e. 6 weeks) after bilateral ovariectomy with or without hysterectomy
  * Women of childbearing potential must have a negative serum pregnancy test performed within 7 days before the first dose of study drug.
  * Continuous and correct application of a contraception method with a Pearl Index of <1% (e.g. implants, depots, oral contraceptives, intrauterine device - IUD) from time point of signing the informed consent until 30 days after the last dose of study drug.

Note: At present, it is not known whether the effectiveness of hormonal contraceptives is reduced by venetoclax. For this reason, women should use a barrier method in addition to hormonal contraceptive methods.

* Sexual abstinence
* Vasectomy of the sexual partner

Inclusion criteria applying for expansion phase (Phase II) only:

• Primary refractory after 1-2 cycles of standard induction chemotherapy (100 to 200 mg/m2 cytarabine over 7-10 days plus anthracycline or mitoxantrone over 3 days or equivalent treatment, e.g. CPX351) or relapsed from first or second CR after 1-2 cycles of standard induction chemotherapy (which must have included cytarabine with an anthracycline or anthracenedione), including relapse after allogeneic stem cell transplantation

Note: Primary refractory disease is defined by either ≥ 20% myeloid blasts on early response assessment around day 15 after start of the most recent induction, or by ≥ 5% myeloid blasts after blood recovery after start of the most recent induction, respectively.

Exclusion Criteria:

* Acute promyelocytic leukemia (AML M3)
* CNS involvement or subjects with extramedullary disease only
* Known hypersensitivity to excipients of the preparation or any agent given in association with this study including cytarabine or mitoxantrone
* Intended hematopoietic stem cell transplantation planned as early conditioning from aplasia without previous blood count recovery
* Cumulative previous exposure to anthracyclines of >410 mg/m2 doxorubicin equivalents
* Acute GVHD ≥ grade 2, extensive chronic GVHD or requiring systemic immunosuppressive therapy within 2 weeks prior to start of study treatment
* HIV infection (due to potential drug-drug interactions between antiretroviral medications and venetoclax, as well as anticipated venetoclax mechanism-based lymphopenia that may potentially increase the risk of opportunistic infections).
* Inability to swallow oral medications
* Any malabsorption condition
* Cardiovascular disability status of New York Heart Association (NYHA) Class ≥ 2.

Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.

* Chronic respiratory disease that requires continuous oxygen use.
* White blood cell count > 25 × 109/L. Note: Hydroxyurea is permitted to meet this criterion.
* AML relapse treatment with any investigational or commercial drug within 14 days before enrolment. Hydroxyurea is allowed until enrolment to control peripheral WBC counts. Toxic effects of previous investigational drug treatment have to recover to Grade <2.
* Substance abuse, medical, psychological, or social conditions that may interfere with the subject's cooperation with the requirements of the trial or evaluation of the study results
* Acute non-hematologic toxicities from any prior anti-leukemia therapy or from previous investigational drugs that have not resolved to Grade <2 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Evens (CTCAE), Version 5.0
* Pregnant or breastfeeding women. Breastfeeding has to be discontinued before onset of and during treatment and should be discontinued for at least 3 months after end of treatment.
* History of active or chronic infectious hepatitis unless serology demonstrates clearance of infection (Occult or prior hepatitis B virus (HBV) infection (defined as negative hepatitis B surface antigen and positive total hepatitis B core antibody) may be included if HBV DNA is undetectable, provided that they are willing to undergo monthly DNA testing. Patients who have protective titers of hepatitis B surface antibody after vaccination or prior but cured hepatitis B are eligible. Patients positive for hepatitis C virus antibody are eligible provided PCR is negative for HCV RNA.)
* History of clinically significant liver cirrhosis (e.g., Child-Pugh class B and C).
* Live-virus vaccines given within 28 days prior to the initiation of study treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (= recommended phase II dose) of cytarabine in combination with venetoclax plus mitoxantrone | appr. 9 months
  number of dose limiting toxicities related to venetoclax per cohort
CR/CRi rate | appr. 12 months
  preliminary efficacy of venetoclax in combination with increasing cytarabine doses plus fixed dose mitoxantrone

SECONDARY OUTCOMES:
remission | appr. 48 months
  Duration of Remission and Depth of remission (MRD)
Relapse | appr. 48 months
  Cumulative incidence of relapse
Relapse-free survival | appr. 48 months
  number of participants alive without relapse
Mortality | appr. 48 months
  Early mortality (within 14 and 30 days)
Proportion of allogeneic stem cell transplantation | appr. 48 months
  number of allogeneic stem cell transplantation following response
incidence and severity of adverse Events [safety and tolerability] | appr. 48 months
  number and grade of Adverse Events assessed by CTCAE v5.0
Overall survival | appr. 48 months
  number of patients alive

OTHER OUTCOMES:
Identification of biomarkers predicting CR/CRi achievement | appr. 48 months
  Baseline samples from all patients with be sequenced for genes which have been associated with response to venetoclax treatment. The panel will include TP53, WT1, PDGFRB, ASXL1, and EZH2. Testing for additional markers may be added triggered by new scientific evidence.
clonal architecture of hematopoiesis | appr. 48 months
  We will test for changes of the clonal architecture of hematopoiesis during therapy and maintenance treatment. This will be done by NGS using a gene panel including TP53, DNMT3A, ASXL1, TET2, JAK2, RUNX1, SF3B1, and EZH2.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Röllig, Prof. (MD), Principal Investigator — Technische Universität Dresden (TUD)
Locations (12):
- Germany (12):
  - Klinikum Augsburg, Medizinische Klinik II, Augsburg
  - Klinikum Chemnitz, Krankenhaus Küchwald, Klinik für Innere Medizin III, Chemnitz
  - Universitätsklinikum Dresden, Medizinische Klinik I, Dresden
  - Universitätsklinikum Essen; Zentrum für Innere Medizin, Essen
  - Universitätsklinikum Frankfurt am Main, Medizinische Klinik II, Frankfurt am Main
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Klinik für Innere Medizin II, Kiel
  - Universitätsklinikum Marburg, Marburg
  - Rotkreuzklinikum München, III. Medizinische Abteilung-Hämatologie und Onkologie, München
  - Universitätsklinikum Münster, Medizinische Klinik A, Münster
  - Klinikum Nürnberg Nord, Klinik für Innere Medizin 5, Nuremberg
  - Robert-Bosch-Krankenhaus Hämatologie, Onkologie und Palliativmedizin, Stuttgart
  - Universitätsklinikum Würzburg, Comprehensive Cancer Center Mainfranken, Würzburg